CLINICAL TRIAL: NCT06925126
Title: Exosome-based Scoring Model for Post-treatment Surveillance of Recurrence in Ovarian Cancer
Brief Title: Exosome-based Recurrence Score for Post-Treatment Ovarian Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaohua Wu MD [zzhong], Director of Gynecological Oncology, Fudan University
Other Study IDs: 2501-Exp131
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Cohort
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — This is an observational cohort study with no planned interventions. Participants will be followed over multiple time points to evaluate treatment outcomes based on the standard care process.

SUMMARY:
The goal of this observational study is to develop an exosome-based scoring model for post-treatment surveillance of recurrence in ovarian cancer. The main questions it aims to answer are:

1. Does this model have the potential for ovarian cancer recurrence monitoring?
2. Can this model demonstrate superior performance to CA125 for ovarian cancer recurrence monitoring?

Participants will :

1. Provide serial blood samples at predefined times
2. Undergo standardized imaging and clinical assessments during follow-up visits

DETAILED DESCRIPTION:
Ovarian cancer is the most lethal gynecologic malignancy with the lowest survival rate among the three major gynecological malignancies. Over 70% of ovarian cancer patients experience recurrence within three years after initial treatment, making treatment response prediction and recurrence monitoring during treatment phases and follow-up visits particularly crucial. CA125 remains the primary recommended biomarker for ovarian cancer recurrence surveillance in current national and international guidelines, while its suboptimal performance necessitates further improvements.

Clinical trial data demonstrated that an exosome-based scoring model, Ovarian Cancer Score (OCS), outperformed CA125 in sensitivity for detecting FIGO stage I ovarian cancer. Notably, OCS results correlated well with FIGO stage and demonstrated improved sensitivity over CA125, particularly in early-stage ovarian cancer, suggesting its potential for recurrence surveillance. This study proposes to develop and validate a new exosome-based scoring model for post-treatment surveillance of recurrence in ovarian cancer, aiming to explore the potential of exosomal biomarkers in cancer recurrence monitoring and ultimately provide clinicians with an effective surveillance tool for ovarian cancer recurrence management.

The study consists of two stages and plans to prospectively enroll 200 patients with epithelial ovarian cancers. In stage I, enrolled patients will be categorized into relapse and non-relapse groups based on their imaging-confirmed recurrence status. Serum exosomal protein profiles obatined from their blood samples will be used for model development. In stage II, patients in the relapse group will undergo standard clinical management with follow-up visits every 3 months. Serum exosomal protein profiles obatined from them will be used for model validation. Overall, blood samples will be collected at enrollment (baseline), after surgery prior to adjuvant chemotherapy (if applicable), during adjuvant chemotherapy or systemic chemotherapy, after adjuvant chemotherapy prior to follow-up visits, and at several time points during follow-up visits. Follow-up visits will continue until either patients experience an ovarian cancer recurrence or the predetermined endpoint of follow-up visits (18 months) is reached. In stage I, logistic regression model will be used to draw a ROC curve and the Youden index will be used to select the most suitable cutoff value. In stage II, sensitivity, specificity, PPV and NPV will be calculated based on results of the model and imaging-confirmed recurrence status. All data will be processed via SPSS 23.0, GraphPad PRISM version 8.0, and R version 4.4.0.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years
* Pathologic confirmed stage I-IV epithelial ovarian cancer, with ≤2 prior lines of therapy (maintenance therapy is not counted as a line of treatment), platinum-sensitive recurrence (achieved complete/partial response [CR/PR] after last platinum-based chemotherapy, with a platinum-free interval >6 months), and radiologically confirmed recurrent disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* A life expectancy of at least 6 months
* Written informed consent

Exclusion Criteria:

* Patients with non-epithelial tumors
* Patients with history of other malignancies within the past 5 years (except completely resected basal cell carcinoma or squamous cell carcinoma of the skin)
* Women who are pregnant, lactating, or intend to become pregnant during the study period
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer affects only biological females, as ovaries are part of the female reproductive system. Thus, research focuses on this population to ensure findings are relevant and applicable to those at risk.
Study Population: Patients with recurrent epithelial ovarian cancer who treated in the Fudan University Shanghai Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | From the end of adjuvant threapy to the end of follow-up visits at 18 months
  The length of time from the date of the end of adjuvant threapy to the date of the first loco-regional or systemic recurrence

IPD SHARING:
Plan to Share IPD: Undecided